CLINICAL TRIAL: NCT00229151
Title: Sleep Deprivation and Three Days Sleep Phase Advancement as Treatment for Bipolar Depression.
Brief Title: Sleep Deprivation and Advancement of Sleep Period as Treatment for Bipolar Depression.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruiting problems
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2005.1.depr
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep deprivation (Experimental): Sleep deprivation and sleep phase advancement
  Interventions: Behavioral: Sleep deprivation and sleep phase advancement
- usual treatment (Active Comparator)
  Interventions: Other: usual treatment

INTERVENTIONS:
Behavioral: Sleep deprivation and sleep phase advancement — Total sleep deprivation from 0800 to 1700 next day, and three day sleep phase advancement following sleep deprivation.
  Arms: Sleep deprivation
Other: usual treatment — Treatment as usual in the psychiatric ward. Patients in this group will be offered treatment with sleep deprivation and sleep phase advancement after five weeks if they still meet inclusion criteria
  Arms: usual treatment

SUMMARY:
The purpose of this study is to determine if sleep deprivation and sleep phase advancement is effective treatment of bipolar patients in a depressive phase.

DETAILED DESCRIPTION:
Background: The onset of therapeutic action for most anti-depressive treatments is usually two weeks. During this period patients suffer from great symptomatic distress. Treatment options that are effective in this period is therefore of interest for psychiatric wards.

Aim: To explore if sleep deprivation and three days sleep phase advancement is effective treatment for inpatients with bipolar disorder in a depressive phase.

Method: A randomized controlled trial with 24 patients diagnosed with bipolar disorder. Patients will be randomized to treatment as usual in an psychiatric ward, or sleep deprivation and three days sleep phase advancement. Patients in the treatment as usual group will be offered treatment with sleep deprivation and sleep phase advancement after five weeks if they still meet inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder, depressive phase

Exclusion Criteria:

* substance abuse, psychotic symptoms, suicidal intentions, active mania/hypomania.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Scores on rating scales for depression and symptom severity. | one month

SECONDARY OUTCOMES:
Scores on rating scales for anxiety, mania, cognitive processing, and sleep quality. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Morken, PhD MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Institute of Neuroscience, Trondheim, Norway